CLINICAL TRIAL: NCT04686656
Title: A Randomized Controlled Trial Comparing Nasal With Buccal Oxygen Administration for Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration
Brief Title: Nasal Versus Buccal Oxygen Administration for Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: tayfun1
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-12

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal oxygen supplementation group (Active Comparator): supplemental oxygen will be administered with nasal cannula
  Interventions: Other: nasal oxygen
- buccal oxygen supplementation group (Active Comparator): supplemental oxygen will be administered with Ring-Adair-Elwyn (RAE) tube
  Interventions: Other: buccal oxygen

INTERVENTIONS:
Other: nasal oxygen — Nasal cannula will be placed by the anesthesiologist. 6 l/ min of supplemental oxygen will be administered with nasal cannula.
  Arms: nasal oxygen supplementation group
Other: buccal oxygen — Ring-adair-elwyn (RAE) tube will be placed by the anesthesiologist. 6 l/ min of supplemental oxygen will be administered with RAE tube.
  Arms: buccal oxygen supplementation group

SUMMARY:
The purpose of this study is to compare to nasal and buccal oxygen administration in patients undergoing Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration .

DETAILED DESCRIPTION:
Anesthesia for Endobronchial Ultrasound (EBUS) may be range from routine bronchoscopy sedation to general anesthesia. During sedation to EBUS increased duration of anesthesia and sedative dosing put patients at increased risk for hypoxic events. To avoid this, oxygen supplementation is mandatory. There are different techniques for oxygen supplementation during the procedure. At this study we will compare to nasal and buccal oxygen supplementations during EBUS.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years of age
* body mass index (BMI) between 20 and 30
* American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* congestive heart failure
* ischemic heart disease
* increased intracranial pressure
* known allergy or contraindication to study drugs (propofol, fentanyl, or midazolam)
* an anatomical feature precluding adequate positioning of the buccal device.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
hypoxia-related interruptions | 30 minutes
  the number of hypoxia-related interruptions

SECONDARY OUTCOMES:
duration of procedure | 30 minutes
  Duration of procedure will be defined in minute as the time from starting to insert EBUS device until the time to remove the device
use of propofol | 30 minutes
  The use of amount of propofol will be noted during the procedure.
use of fentanyl | 30 minutes
  The use of amount of fentanyl will be noted during the procedure.
satisfaction of pulmonary specialist | 30 minutes
  satisfaction of pulmonary specialist will be evaluated by 4-points Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: tayfun sugur, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Researching Hospital, Antalya, Turkey (Türkiye)